CLINICAL TRIAL: NCT05549895
Title: Effect of Intrathecal Dexamethasone on Intra-operative Hemodynamic in Elderly Patients Undergoing Urologic Endoscopic Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dalia Mohamed Abbas, Assistant lecture, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Intrathecal Dexamethasone
Record Dates: First submitted 2022-05-27; First posted 2022-09-22 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Dexamethasone; Urologic Endoscopic Surgery
MeSH Terms: interventions — Dexamethasone; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug arm (Experimental): 45 patients will receive 8mg dexamethasone in addition to bupivacaine intrathecally .
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine Hydrochloride
- control arm (Other): 45 patients will receive only bupivacaine intrathecally as a control group.
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Dexamethasone — 8 mg intrathecally
  Arms: Drug arm
Drug: Bupivacaine Hydrochloride — 0.5 % intrathecally

SUMMARY:
Correction of Post-spinal anesthesia hypotension by fluids pose the risk of volume overload or compromising cardiac conditions. Intravenous Dexamethasone in some studies is used to treat conditions manifested by decrease of peripheral vascular resistance Many advantages were investigated for the addition of dexamethasone to bupivacaine in spinal anesthesia as prolongation of anesthesia time, postoperative analgesia and prophylaxis for shivering.

In this study the investigators will investigate the ability of dexamethasone to blunt post-spinal anesthesia hypotension in elderly patients undergoing urological endoscopic surgery, and hence, if it decreases amount of fluids and dose of vasoactive drugs.

DETAILED DESCRIPTION:
Spinal anesthesia is the most consistent block for lower abdomen and lower limb surgery. Spinal anesthesia avoids the risks of general anesthesia such as aspiration of gastric contents and difficulty with airway management.

Post-spinal anesthesia hypotension in elderly patients is challenging. Correction of Post-spinal anesthesia hypotension by fluids either colloids or crystalloids or by vasoconstrictors pose the risk of volume overload or compromising cardiac conditions. Intravenous Dexamethasone in some studies is used to treat conditions manifested by decrease of peripheral vascular resistance.

Many advantages were investigated for the addition of dexamethasone to bupivacaine in spinal anesthesia as prolongation of anesthesia time, postoperative analgesia and prophylaxis for shivering. Avoidance of complications of opioids is a great issue as, postoperative nausea, vomiting, respiratory depression, urinary retention, prolonged hospital stay and immunosuppression.

In this study the investigators will investigate the ability of dexamethasone to blunt post-spinal anesthesia hypotension in elderly patients undergoing urological endoscopic surgery, and hence, if it decreases amount of fluids and dose of vasoactive drugs.

ELIGIBILITY:
Inclusion Criteria:

* Age: > 60 years old
* Gender: Males and females
* ASA grade I - II - III
* Patients undergoing elective endoscopic urological procedures.

Exclusion Criteria:

* Patient refusal.
* Suspected massive bleeding.
* Transition to open abdominal surgery

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Total amount of fluids | intraoperative
  Total amount of fluids needed to maintain mean blood pressure more than 65 mmHg
Total amount of vasoactive drugs | Intraoperative
  Total amount of vasoactive drugs needed to maintain mean blood pressure more than 65 mmHg

SECONDARY OUTCOMES:
Blood pressure | Intraoperative and up to 1hour postoperative
  systolic and diastolic blood pressure and mean arterial blood pressure.
Post-operative VAS score of pain assessment. | Up to one hour postoperative
  Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
Post-operative shivering. | Up to 6 hours postoperatively.
  shivering of the patient
Post-operative nausea and vomiting. | Up to 6 hours postoperatively.
  The presence of nausea or vomiting 6 hours post operatively
Post dural puncture headache. | Up to 2 days postoperative
  headache during 2 days postoperative and detection of severity and response to treatment